CLINICAL TRIAL: NCT05361811
Title: Acceptance and Commitment Therapy for Caregivers of Children With a RASopathy: An Internal Pilot Feasibility Study and Follow-up Phase III Randomized Controlled Trial
Brief Title: Acceptance and Commitment Therapy for Caregivers of Children With a RASopathy: An Internal Pilot Feasibility Study and Follow-up Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10000657; 000657-C
Record Dates: First submitted 2022-05-03; First posted 2022-05-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Neurofibromatosis 1; Noonan Syndrome; Legius Syndrome; Cardiofaciocutaneous Syndrome; Costello Syndrome
Keywords: Parenting; Stress; Parent; Therapist; Coach; virtual; Quality of Life; Genetic Condition; Rare
MeSH Terms: conditions — Neurofibromatosis 1; Noonan Syndrome; Legius syndrome; Cardiofaciocutaneous syndrome; Costello Syndrome; Genetic Diseases, Inborn | interventions — Waiting Lists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1/Internal Pilot (Experimental): Participants will begin their 1-week baseline EMA data collection period and then take part in intervention procedures immediately after enrollment to assess feasibility and acceptability.
  Interventions: Behavioral: ACT Intervention
- 2/Immediate Intervention (Active Comparator): Participants will begin their 1-week baseline EMA data collection period immediately after randomization and will begin receiving the 8-week intervention at the end of this week/beginning of the next week (depending on participant schedule).
  Interventions: Behavioral: ACT Intervention
- 3/Waitlist Control (Active Comparator): After an initial 1-week baseline period for EMA data collection and 8 weeks of maintaining their usual routine (wait list period), participants will begin receiving the 8-week intervention.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Waitlist — 8 weeks of maintaining usual routine followed by 8-week intervention that emphasizes mindfulness, acceptance, perspective taking, and values-based actions.
  Arms: 3/Waitlist Control
Behavioral: ACT Intervention — 8-week intervention that emphasizes mindfulness, acceptance, perspective taking, and values-based actions.
  Arms: 1/Internal Pilot; 2/Immediate Intervention

SUMMARY:
Background:

RASopathies are a group of genetic diseases that affect a child s development. They cause physical, cognitive, and behavioral symptoms. Caring for a child with a RASopathy can be stressful. Acceptance and Commitment Therapy (ACT) is a therapy that helps people become more aware and accepting of difficult thoughts and feelings. ACT has been found to be helpful for parents with high parenting stress.

Objective:

To find out if Acceptance and Commitment Therapy (ACT) can help caregivers of children with a RASopathy better cope with parenting stress.

Eligibility:

People aged 18 years or older who care for a child (younger than 18 years) with a RASopathy. The child must live with the caregiver at least 50% of the time.

Design:

The study is fully remote. Participants need a mobile device that can play audio and video and connect to the internet. They can borrow an iPod if needed.

Participants will download a free app called MetricWire. They will use this app to watch videos and answer questions.

The first 8 participants will be in a pilot study. They will receive the ACT intervention starting the first week after they begin the study.

After the pilot study, we will start a new phase called the randomized trial. In this phase, participants will have a 50-50 chance of being in the group that will start the intervention right away or the group that will start the intervention after about 2 months.

Participants will fill out surveys on 5 random days each week. These surveys have 7 questions and take about 2 minutes. They will also fill out 3 longer questionnaires: once before ACT begins, once just after the 8-week study period, and once about 3 months later. Questions will cover topics including:

Parenting stress

Life satisfaction

Self-compassion

Uncomfortable feelings and thoughts

Mindfulness

Participants will take part in an 8-week ACT intervention. They will have one 75-minute session with an ACT coach in the first week.

Participants will watch 9- to 17-minute videos each week. The videos talk about how to practice ACT techniques to cope with parenting stress.

Participants will have 20- to 30-minute coaching sessions in weeks 3 and 6. The coach will help them practice exercises and work through any problems.

DETAILED DESCRIPTION:
Background:

* RASopathies are a group of neurodevelopmental genetic conditions caused by mutations affecting components within the RAS-map kinase (RAS-MAPK) cellular signaling pathway.
* Caregivers of children with a RASopathy are faced with numerous challenges related to the physical, cognitive, and behavioral symptoms associated with their child s condition.
* The use of virtual interventions has been increasing over the past decade, which increase accessibility and are especially critical during times of physical distancing, such as due to COVID-19.
* Similarly, Ecological Momentary Assessments (EMA) are being utilized more frequently in order to maximize ecological validity of results and minimize recall bias.
* To our knowledge, no psychological interventions have been investigated targeting parenting stress among caregivers of a child with a RASopathy.

Primary Objectives:

* Internal Pilot Study: To assess the feasibility (e.g., enrollment and attrition) and acceptability (e.g., satisfaction) of an Acceptance and Commitment Therapy (ACT) coping intervention on parenting stress for caregivers of a child with a RASopathy
* Randomized Controlled Trial (RCT): To compare Parental Stress Scale (PSS) changes from baseline to 8 weeks between the Immediate Intervention Arm and the Waitlist Control Arm

Eligibility:

* Caregiver (parent or legal guardian) of a child (< 18 years) residing with them at least 50% of the time who has a diagnosis of RASopathy syndrome including NF1, Noonan Syndrome, Legius Syndrome, Cardiofaciocutaneous (CFC) syndrome, and Costello Syndrome, or another RASopathy
* Access to necessary resources for participating in a technology-based intervention (i.e., computer, smartphone, internet access) or be willing to use an iPod provided by the study team
* Must score a 15 or higher total score on modified questions from the PSS to indicate at least a moderate level of parenting stress
* Ability to read and speak English

Design:

* This is an 8-week psychological intervention study that has two phases: the first, an internal pilot study, will enroll an initial, small cohort of caregivers (n = 8), all of whom will participate in the ACT intervention. (COMPLETE)
* Due to the success of the internal pilot study (with specific benchmarks met), the second phase of this study will be an RCT comparing participants who receive the intervention immediately (Immediate Intervention Arm) with those in a control group (Waitlist Control Arm). Participants randomized to the Waitlist Control Arm will cross over to receive the intervention after the waitlist period.
* The intervention for the RCT phase involves a baseline 90-minute coaching session and two follow-up coaching sessions with a therapist over video chat, followed by weekly prerecorded video modules that the participants can view at their convenience over the following 8 weeks.
* Participants will complete measures of parenting stress, mindfulness, psychological flexibility, self-compassion, and perceptions of child well-being at baseline, the 8-week post-intervention assessment, and a 3-month follow-up assessment. Additionally, the study will use EMA whereby questions will be sent electronically at random times and days (once a day at varying times on 5 days a week) during weeks 0-8 (the first week will serve as baseline data for comparison) for the Immediate Intervention Arm and weeks 0-18 for the Waitlist Control Arm using the Catalyst mobile application by MetricWire software.
* We plan to enroll 8 participants in the internal pilot phase and 56 participants in the RCT phase to account for the potential attrition of two caregivers from the intervention, for a total accrual target of 64 evaluable participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ability to understand and the willingness to sign a written informed consent document
* Ability to read and speak English
* Age >= 18 years
* Caregiver (defined as parent or legal guardian) of a child (< 18 years) with a diagnosis of a RASopathy syndrome including NF1, Noonan Syndrome, Legius Syndrome, CFC, and Costello Syndrome, or another RASopathy
* The participant s child with a RASopathy must live with them at least 50% of the time
* Access to necessary resources for participating in a technology-based intervention (i.e., computer, smartphone, internet access) or be willing to use an iPod provided by study team.
* Must score a 15 or higher total score on modified questions from the Parental Stress Scale (PSS), indicating endorsement of the midpoint response on average and thus a moderate level of parenting stress.
* Caregiver must not be participating in or planning to participate in psychosocial intervention primarily targeting parenting stress over the duration of the study. Caregivers are able to receive interventions for other mental health concerns as long as parenting stress is not the main focus of treatment.

EXCLUSION CRITERIA:

* Another caregiver in the same household is participating in this protocol. If two caregivers in the same household want to participate, we will inform them that one can enroll on the protocol and the other can receive the intervention materials (e.g., parent workbook, audio recordings) to practice on their own. The reason for this is that parents participating with their partner may interact with the intervention differently and have more direct support than other participants. We will collect data on how many caregivers live in the household and how often the second parent engaged with the parent workbook and audio recordings in our pre and post study questionnaires.
* Uncontrolled psychiatric illness, cognitive impairments, or other circumstance as judged by the Principal Investigator, a licensed psychologist, that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility & Acceptability | 9 weeks
  Feasibility defined by compliance with viewing >50% of the weekly videos (proposed target rate of 5 out of 8 videos watched; must watch at least 80% of each video), and 70% of participants attending both coaching sessions 2 and 3. Acceptability defined by descriptive data per caregiver reports of satisfaction on the Study Satisfaction survey (mean of questions 1-7 and 9).
Changes in PSS | 9 weeks
  RCT: Mean scores on the Parental Stress Scale (PSS) will be compared from pre- to post-intervention (baseline to 8 weeks between the immediate intervention arm and the wait list control arm.

SECONDARY OUTCOMES:
To examine the feasibility of ecological momentary assessment methods to assess patterns of parenting stress levels over time | 21 weeks
  Feasibility defined by compliance with daily surveys (target rate of 30 out of 40 surveys (75%) completed on average by each participant). Acceptability defined by post-intervention participant reports of satisfaction with completing daily EMA ratings on the Study Satisfaction survey.
To examine changes on caregiver-completed measures of psychological flexibility, self-compassion, experiential avoidance, depression, and perceptions of child affect from pre- to post-intervention | 21 weeks
  We will examine pre- to post-intervention changes in scores on measures of psychological flexibility (MPFI-SF), self-compassion (SCS-SF), experiential avoidance (BEAQ), depression (PROMIS Depression 8a) and child affect (PROMIS Positive Affect Scale).
To determine whether psychological flexibility mediates the relationship between treatment group and parenting stress | 21 weeks
  We will look for a significant indirect association between treatment arm assignment and pre- to post-intervention PSS changes via psychological flexibility as measured by the BEAQ.

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000657-C.html